CLINICAL TRIAL: NCT05312294
Title: Multicenter, Double-blind, Comparative, Randomized Tolerability, Safety and Immunogenicity Trial of the Flu-M® Inactivated Vaccine in Volunteers Aged 18 to 60 Years
Brief Title: Tolerability, Safety and Immunogenicity Trial of the Flu-M® Inactivated Vaccine in Volunteers Aged 18 to 60 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FLM-03-2020
Record Dates: First submitted 2022-03-17; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Influenza; Flu, Human
Keywords: Influenza; Flu; Vaccine; FLU-M; SPbSRIVS
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLU-M w/o/p (Experimental): Volunteers were vaccinated with a single dose of the Flu-M vaccine (without preservative) intramuscularly in a dose of 0.5 mL.
  Interventions: Biological: Flu-M [inactivated split influenza vaccine] without preservative
- FLU-M w/p (Experimental): Volunteers were vaccinated with a single dose of the Flu-M vaccine (with preservative) intramuscularly in a dose of 0.5 mL.
  Interventions: Biological: Flu-M [inactivated split influenza vaccine] with preservative

INTERVENTIONS:
Biological: Flu-M [inactivated split influenza vaccine] without preservative — Solution for intramuscular injection, 0.5 ml
  Arms: FLU-M w/o/p
Biological: Flu-M [inactivated split influenza vaccine] with preservative — Solution for intramuscular injection, 0.5 ml
  Arms: FLU-M w/p

SUMMARY:
Comparative assessment of the tolerability, safety, and immunogenicity of the Flu-M® Inactivated Split Influenza Vaccine (without preservative) and the Flu-M® vaccine (with preservative) in volunteers aged between 18 and 60

DETAILED DESCRIPTION:
1. Assessment of the tolerability and safety of the Flu-M® inactivated split influenza vaccine (without preservative) and Flu-M® (with preservative).
2. Assessment of the immunogenicity of the Flu-M® inactivated split influenza vaccine (with preservative) and Flu-M® (without preservative).

Single administration of the trial products. Duration of follow-up - 28+3 (outpatient visit) and Long-term follow-up - 180±3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers (men and women) aged 18-60 years;
2. Written informed consent of volunteers to participate in the clinical trial;
3. Volunteers able to fulfill requirements of the Protocol (i.e. fill out the patient's diary, come to follow-up visits);
4. For fertile women - a negative result of the pregnancy test and consent to observe adequate methods of contraception during the trial and at least two months after vaccination
5. For fertile men - consent to observe adequate methods of contraception during the trial and at least two months after vaccination, except for men after vasectomy with documented azoospermia, and their sexual partners should use methods of contraception that ensure more than 90% reliability or be incapable of conception after a surgical sterilization or have a natural menopause for at least 2 years.

Exclusion Criteria:

1. History of influenza/ARVI or previous influenza vaccination during 6 months before the trial;
2. Positive result of the SARS-CoV-2 test;
3. A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination);
4. Allergic reactions to vaccine components or any previous vaccination;
5. History of allergic reaction to chicken protein;
6. Guillain-Barré syndrome (acute polyneuropathy) in the medical history;
7. Previous vaccination with rabies vaccines less than 2 months before immunization or scheduled vaccination with rabies vaccines within 1 month after immunization with the trial vaccines;
8. Use of any vaccines within 1 month before the vaccination, excluding vaccines according to the National Calendar of Preventive Vaccination, including for epidemic reasons;
9. History of leukemia, cancer, autoimmune diseases;
10. (Positive blood test results for HIV, syphilis, hepatitis B/C;
11. Volunteers who received immunoglobulin or blood products or had a blood transfusion during the last three months before the trial;
12. History of long-term use (more than 14 days) of immunosuppressants or immunomodulatory drugs for six months before the trial;
13. History of any confirmed or suspected immunosuppressive or immunodeficiency condition;
14. History of chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, the gastrointestinal tract, liver, kidneys, hematopoietic or immune systems, mental disease in the acute stage or in the decompensation stage (recovery less than 4 weeks before vaccination);
15. Diabetes mellitus, thyrotoxicosis or other diseases of the endocrine system;
16. History of eczema;
17. Treatment with glucocorticosteroids, including in small doses, as well as local use of drugs containing steroids (> 10 mg of prednisolone or its equivalent for more than 14 days before the screening);
18. Tuberculosis, neurological or mental disorders, a convulsive syndrome, including in the past medical history;
19. History of acute infectious diseases (recovery less than 4 weeks before vaccination);
20. Consumption of more than 10 units of alcohol per week or history of alcohol addiction, drug addiction or abuse of pharmaceutical products;
21. Smoking of more than 10 cigarettes per day;
22. Participation in another clinical trial during the last 3 months;
23. Pregnancy or lactation;
24. Coagulopathy, including hemophilia;
25. Taking aspirin or other antiplatelet agents in high doses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 654 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline geometric mean titer ratio of antibodies for each virus strain (GMT (Flu-M w/p) / GMT (Flu-M w/o/p) at 6 months | days 0-180
  The upper limit of bilateral 95% CI for the GMT ratio (GMT (Flu-M w/p) / GMT (Flu-M w/o/p) should not exceed 1.5
Change from baseline the difference between seroconversion rates (seroconversion rate Flu-M w/p - seroconversion rate Flu-M w/o/p) at 6 months | days 0-180
  The upper limit of bilateral 95% CI for the difference between seroconversion rates (seroconversion rate Flu-M w/p - seroconversion rate Flu-M w/o/p) should not exceed 10%

SECONDARY OUTCOMES:
Geometric mean titer of antibodies for each virus strain (A (H1N1), A (H3N2) and B) | days 0,28,180
  Specific anti-influenza antibodies were determined using haemagglutination inhibition assay (HI assay)
Seroconversion rate for each virus strain (A (H1N1), A (H3N2) and B) | days 0,28,180
Seroconversion factor for each virus strain (A (H1N1), A (H3N2) and B) | days 0,28,180
Seroprotection rate for each virus strain (A (H1N1), A (H3N2) and B) | days 0,28,180
Incidence, severity, and duration of influenza or ARVI during 6 months after vaccination | days 1-180
Incidence of adverse events (AEs) | days 1-180
Incidence of serious adverse events (SAEs) | days 1-180
Number of patients with abnormal results of blood pressure (BP) | days 0,1,7,28,180
  BP measurements include the systolic and diastolic blood pressure.BP is measured on the brachial artery according to the Korotkoff method using a certified sphygmomanometer or tonometer. It is also allowed to use a certified electronic tonometer for measuring.
Number of patients with abnormal results of heart rate (HR) | days 0,1,7,28,180
  The HR is measured during auscultation of the heart in parallel with determining the pulse rate on the radial artery (or on the carotid artery in case of weak pulsation in the radial artery) for a minute while sitting.
Number of patients with abnormal results of respiratory rate (RR) | days 0,1,7,28,180
  The RR is measured for a minute at rest in the sitting position, by registering the breathing movements of the chest or abdominal wall.
Number of patients with abnormal results of body temperature (>37 °С) | days 0,1,7,28,180
  Body temperature (°C) is measured with a mercury or digital thermometer in the armpit for at least 5 minutes or with a non-contact infrared digital thermometer.
Number of patients with abnormal results of physical examination | days 0,1,7,28,180
  Physical examination of volunteers includes an interview, discovery of complaints and symptoms, when required, palpation, auscultation, percussion.
Number of patients with abnormal results of neurological status | days 0,7,28
  Assessment of:
  * Cranial nerve function
  * Motor sphere
  * Reflex sphere
  * Sensitive sphere
  * Coordination sphere
  * Pelvic functions
  * Higher mental functions
Determination of total IgE | days 0,7,28
Number of patients with abnormal results of electrocardiography (ECG) | days 0,7
  2-lead electrocardiography (ECG). Assessment of: PQ, QT,QTc intervals, QRS complex

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - State Autonomous Health Institution "Engels City Clinical Hospital No1", Engel's
  - Limited Liability Company "Professorskaya Clinica", Perm
  - Limited Liability Company "Clinika Zvezdnaya", Saint Petersburg
  - Limited Liability Company "MEDICINSKAYA CLINIKA", Saint Petersburg
  - Limited Liability Company "PeterClinic", Saint Petersburg
  - Limited Liability Company "Scientific Research Center Eco-Safety", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "State Polyclinic No. 117", Saint Petersburg
  - Limited Liability Company "Medical Center Diagnostics and Prevention Plus", Yaroslavl